CLINICAL TRIAL: NCT01221545
Title: A Randomised, Single-Blind, Placebo-Controlled, Single-Centre Phase I Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics After High Single Ascending Oral Supratherapeutic Doses of AZD1656 in Male Type 2 Diabetes Mellitus (T2DM) Patients
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics After High Single Ascending Oral Doses of AZD1656 in T2DM Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Eva Johnsson MSD, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: D1020C00044
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — AZD1656

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - AZD1656 (Experimental): AZD1656
  Interventions: Drug: AZD1656
- B - Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — 3 escalating dose levels are planned. Administration of the escalating doses of AZD1656 will be based on review of available safety from the previous dose.
  Arms: A - AZD1656
Drug: Placebo — Placebo
  Arms: B - Placebo

SUMMARY:
The purpose of this study is to investigate safety and tolerability after high Single Ascending Oral Doses of AZD1656.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study specific procedures.
* Male, T2DM patients aged 20-60 years
* Treatment with 1 to 2 OADs as Therapy for T2DM for at least 30 days prior to enrollment
* Patients should not have been treated with glitazones within 6 months prior to enrollment
* Male T2DM patients without known cardiovascular disease, with the exception of Grade 1 hypertension without secondary organ involvement (eg. grade 1 HT is allowed if no eye, kidney disease or LVH has been documented).

Exclusion Criteria:

* History of ischemic heart disease , heart failure, stroke, transitory ischemic attack or peripheral vascular disease.
* Prolonged QTcF>450 msec or shortened QTcF<350 msec or family history of long QT syndrome.
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes.
* Systolic BP>159 mmHg or diastolic BP>99 mmHg at screening and on Day-1

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Primary Objective to assess the safety and tolerability of AZD1656, following oral administration of single ascending supratherapeutic doses of AZD1656 to patients with type 2 diabetes mellitus in a fasted state. | From screening until Follow up

SECONDARY OUTCOMES:
Secondary objective to evaluate the pharmacokinetics (AUC, Cmax, t1/2, CL/F) of AZD1656 and its metabolite following oral administration of single ascending supratherapeutic doses of AZD1656 | From pre-dose Day 1 to 48 hours after dose
Secondary objective to evaluate glucose levels and insulin secretion in type 2 diabetes mellitus patients following oral administration of single ascending supratherapeutic doses of AZD1656 | Glucose levels from Day -1 to day 3
Secondary objective to evaluate glucose levels and insulin secretion in type 2 diabetes mellitus patients following oral administration of single ascending supratherapeutic doses of AZD1656 | Insuline secretion from Day -1 to 2.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Morrow, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Research Site, Chula Vista, California, United States